CLINICAL TRIAL: NCT04612400
Title: Whole Body Protein Metabolism of a Whey/EAA Supplement Using Continuous Oral Stable Isotopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 260813
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Stable Isotopes; Validation; Whole-body protein metabolism

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized, crossover pilot study
Who Masked: Participant, Investigator
Masking Description: This will be a double-blinded study. Both SP amounts are dissolved into equal volumes of water so that subjects will not know which amount they are ingesting. Blood samples are coded so that lab staff and investigators will not know which amount of SP was consumed at each visit. Investigators will be unblinded after all samples have been processed and data analysis has taken place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low (Experimental): Low dose (6.3g) EAA/whey protein supplement
  Interventions: Other: Oral amino acid tracer
- High (Experimental): High dose (12.6g) EAA/whey protein supplement
  Interventions: Other: Oral amino acid tracer

INTERVENTIONS:
Other: Oral amino acid tracer — Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.

SUMMARY:
To evaluate the validity of a continuous oral sip-feeding method of stable isotope tracer for the evaluation of whole-body protein metabolism in response to two different doses of an EAA/whey protein supplement (Low=6.3g and High=12.6g). Results will be compared to those previously determined by constant infusion with the same EAA/whey supplement.

DETAILED DESCRIPTION:
This will be a double-blinded, randomized, crossover pilot study to evaluate the validity of a continuous oral sip-feeding of stable isotope tracer method for the evaluation of whole-body protein metabolism. This method will be evaluated using two different amounts of an essential amino acid (EAA) + whey protein supplement on up to six younger, healthy subjects. Stable isotope preparations will be continuously consumed by subjects throughout visits 2 and 3 to enable whole body protein metabolism to be measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-40 years.
* Body weight of ≤ 80kg.

Exclusion Criteria:

* History Chronic kidney disease.
* History of dairy allergy or intolerance.
* History of gastric reduction/bypass surgery.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Center of Translational Research in Aging and Longevity, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Then High Dose: Low dose (6.3g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
- High Dose Then Low Dose: High dose (12.6g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
Period: Overall Study
Arm/Group | Low Dose Then High Dose | High Dose Then Low Dose
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Then High: Low dose (6.3g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
- High Dose Then Low: High dose (12.6g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
- Total: Total of all reporting groups
Arm/Group | Low Dose Then High | High Dose Then Low | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5.3) | 29 (7) | 29 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Whole-body Protein Net Balance
Description: grams of protein per 240 minutes as determined using stable isotope ingestion and blood analysis for said isotopes' concentrations.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Low Dose: Low dose (6.3g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
- High Dose: High dose (12.6g) EAA/whey protein supplement
  Oral amino acid tracer: Whole body protein metabolism response to a dose of the supplement will be measured using a continuous oral sip-feeding (every 10 minutes) method of stable isotope tracer.
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 8 | 8
grams | 6.2 (5.1) | 11.8 (3.9)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT04612400/Prot_SAP_000.pdf